CLINICAL TRIAL: NCT03938909
Title: Ccf mtDNA as a Biomarker in Neurological and Neurodegenerative Diseases
Brief Title: Ccf mtDNA as a Neurodegenerative Biomarker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Stefano Gambardella, Doctor, Principal Investigator, Neuromed IRCCS
Other Study IDs: CGM-03
Record Dates: First submitted 2019-04-16; First posted 2019-05-06 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — CSF, Serum, Plasma, Blood, DNA and RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Multiple Sclerosis: 200 patients and 200 control
  Interventions: Genetic: cif mtDNA biomarker
- Patients with dementia: 100 patients and 100 control
  Interventions: Genetic: cif mtDNA biomarker
- Patients with Parkinson's disease: 50 patients and 50 control
  Interventions: Genetic: cif mtDNA biomarker

INTERVENTIONS:
Genetic: cif mtDNA biomarker — The aim is to evaluate the role of ccf-mtDNA as a specific and early biomarker for different clinical pictures

SUMMARY:
There is a long history of research into body fluid biomarkers in neurodegenerative and neuroinflammatory diseases. However, only a few biomarkers in cerebrospinal fluid (CSF) are being used in clinical practice. One of the most critical factors in biomarker research is the inadequate linkage of biological samples with data from medical records, environmental exposure, lifestyle information and other medically relevant information. In this context the biobanks are an invaluable resource for medical research and, in particular, for the identification of biomarkers. This project aims to enstablish a biobank for Multiple Sclerosis that allow to collect periodically, at each follow up, clinical data, tissues such as blood and cerebrospinal fluid and DNA, RNA, proteins, from patients afferent at the Centre for the Study and Cure of Multiple Sclerosis in Neurological Institute "Neuromed", Pozzilli, Isernia. The samples stored in this biobank are examined by quantization of a potential innovative biomarker focused on the formation of circulating mitochondrial DNA. Fragments of mitochondrial DNA (mtDNA) are released outside the cell and they appear to persist in extracellular ﬂuids as circulating, cell-free, mtDNA (ccf-mtDNA).

This occurs during acute inﬂammation, which anticipates the neurodegenerative process. Thus, an increase in inﬂammatory cells in the affected regions is expected to add on mtDNA release into the CSF. Thus, ccf-mtDNA may represent a powerful biomarker for disease screening and prognosis at early stage, although its biological role may extend to generating the neurobiology of disease.

Aims:

1. Identify a technique that allows to isolate, the mitochondrial DNA circulating from different biological tissues (Droplet Digital PCR, Real Time PCR).
2. Use different technologies to quantify the presence of circulating mitochondrial DNA
3. Use circulating mitochondrial DNA as a biomarker of neurodegenerative and / or neuroinflammatory pathologies.

It is essential to understand the tissue specific origin of circulating mtDNA for both diagnostic and therapeutic considerations. . We believe that our current knowledge on cell free circulating mtDNA is in a rather exploratory phase with a potential for the future to rewrite the pathology of the leading causes of morbidity and mortality such as inflammatory conditions, autoimmune disorders, cancer, heart disease, stroke and injury.

DETAILED DESCRIPTION:
To date, the specific causes of multiple sclerosis (MS) remain uncertain, and in its pathogenesis an interaction between environmental and genetic factors has been implicated leading to inflammation, demyelination and neurodegeneration of the central nervous system (CNS). Epidemiological studies conducted in ethnic groups of families, twins, half sibs and conjugate pairs support a genetic component to this process. The risk for monozygotic twins is 300-times, and for first-degree relatives 20-50-times higher than for an individual in the general population of Northern-European origin with a prevalence rate of 0.1. The transmission patterns observed are not compatible with an autosomal dominant, recessive or X-linked inheritance. MS is a complex trait disorder, defined by several genes, each exerting small effect, and in an interaction with the environment. Phenotypic expressions of MS suggest the involvement of complex mechanisms with features of autoimmunity and neurodegeneration. The currently approved disease modifying drugs are mainly targeted towards the inflammatory components, but exert a limited effect on neurodegeneration in MS. The cognitive impairment can be an early feature of the demyelinating disease process, and in a few cases dementia has been documented in the absence of severe neurological signs. There are some correlation between disease subtype and cognitive impairment: in fact, it is well known that cognitive impairment occurs more frequently and is more severe in patients with progressive rather than in relapsing-remitting MS. Impairment of cognitive domains such as memory, mental processing speed attention and executive function can occur from the early stage of the diseases and tend to worsen over time. Moreover, the underlying pathophysiological mechanisms of the cognitive impairment and neuropsychiatric disorders observed in MS are not fully understood. White matter abnormalities alone cannot fully explain the extent of clinical symptoms in MS, including cognitive impairment. Furthermore, several MRI techniques have shown the involvement of gray matter in MS and the association between gray matter damage, physical disability and cognitive impairment. Therefore, biomarkers that reliably capture the different aspects of disease heterogeneity are needed, and might help to better understand MS disease aetiopathogenesis, diagnosis, and prognosis, to predict response outcome to treatments, and to develop new treatments.

In particular, there is increasing effort to develop molecular diagnostic markers that meet requirements like easy accessibility e.g., from blood, high specificity and sensitivity, low costs and applicability by laboratories with standard equipment. Several blood, plasma, or serum MS biomarkers have been proposed to meet these criteria. In order of this the circulating markers are represented, in addition to the classic serum markers, also by the cells and by free circulating nucleic acids (DNA, RNA). In recent years, among the circulating nucleic acids, a possible role of mitochondrial DNA has emerged as a biomarker in the diagnosis of numerous pathologies.

In humans, mtDNA is significantly smaller when compared with nuclear DNA (16.569bp vs. 3.2 billion bp), and it possesses only 37 genes, among which 13 encode proteins belonging to the respiratory electron transport chain. Unlike nuclear DNA, mtDNA is devoid of protective histones and sophisticated DNA repair mechanisms, which makes it vulnerable to genotoxic stimuli including oxidative stress. In fact, high levels of reactive oxygen species (ROS) are generated around mtDNA during oxidative phosphorylation occurring in mitochondria. Such an oxidative environment contributes to a high susceptibility of mtDNA to mutagenesis. In fact, mtDNA possesses roughly a 10- to 200-fold higher rate of mutagenesis than nuclear DNA under a comparable oxidative stress environment. This may be detrimental for those high-energy-demanding and post-mitotic cells including neurons and myocytes, which are mostly sensitive to altered respiratory chain activity and ROS-mediated damage yielded by mtDNA changes. Such a specific vulnerability of mtDNA determines the occurrence of a detectable amount of mitochondrial DNA fragments, which are released into the bloodstream as circulating, cell-free fragments (ccf-mtDNA). These correspond to double-stranded DNA molecules, which are biologically fragmented into both short (lower than 1 Kb) and long (up to 21 kb) segments. The high rate of mtDNA fragmentation is key in generating ccf-mtDNA, though it remains unclear whether mtDNA is released due to a disruption of the plasma membrane or it is actively extruded from the cell. For instance, oxidative stress or other stimuli can damage cell integrity, while producing apoptosis or necrosis, which in turn lead to mtDNA extrusion from the cell or release into the blood. Nonetheless, even in baseline conditions when the plasma membrane is intact, fragments of mutated mtDNA could be compartmentalized within cytosolic organelles and then released extracellularly. This latter mechanism would guarantee the preservation of mitochondrial function by removing dysfunctional mutated DNA fragments. This is supported by recent work from C. elegans neurons, which expel dysfunctional mitochondria when exposed to neurotoxic stress. Nonetheless, the biological role of ccf-mtDNA and its fragments is still controversial and it needs to be fully understood. In fact, DNA fragments may act as toxic molecules, which in turn impair mitochondrial function and cell membrane, and could also act on cell integrity and tissue repair. This is largely bound to the established, yet double faceted, involvement of mtDNA in innate immunity and inflammation. In fact, similar to bacterial DNA, mtDNA possesses non-methylated CpG sites, which once released in either cytosol or extracellular space behave as damage-associated molecular patterns (DAMPs) to activate innate immunity and inflammation. This occurs via specific biochemical cascades involving the binding of mtDNA to Toll-like receptor 9 (TLR9) and subsequent activation of the stimulator of interferon genes (STING) pathway. These are key in generating inflammatory responses including antimicrobial immunity and neuro-immunological disorders. In fact, DAMPs accumulation activates resident macrophages and fosters tissue infiltration by leukocytes. As for most molecules involved in the immune response, the bulk of evidence concerning the measurement of ccf-mtDNA and its role in physiology and disease stems from studies carried out outside the CNS. In fact, ccf-mtDNA has been analysed in various clinical conditions like neoplasia, trauma, infections, stroke and cardiovascular diseases, where it has been tested as diagnostic and predictive biomarker. Only recently, mtDNA started being evaluated in neurological disorders. In line with the higher resistance of mtDNA to nuclease-dependent degradation compared with nDNA, mtDNA persists as ccf-mtDNA within extracellular ﬂuids including the CSF.

CNS disorders featuring a strong inﬂammatory response are characterized by elevated plasma mtDNA level. In fact, elevated CSF ccf-mtDNA occur in relapsing-remitting (RRMS) and PMS. RRMS is characterized by an acute inﬂammatory response, which precedes neurodegeneration. Thus, the increase in ccf-mtDNA observed in RRMS is a direct consequence of increased activation of inﬂammatory cells. These cells release mtDNA in addition to nDNA, into the CSF. A persistent inflammatory reaction may recruit circulating immune cells while triggering a systemic response through the activation of mtDNA-induced inflammatory pathways. In this way, a vicious circle occurs where inflammatory cytokines and ROS may induce further damage to mitochondria and mtDNA. In this scenario, elevated ccf-mtDNA concentration in MS may reflect early, active inflammatory activity, which eventually culminates in mitochondrial damage, neural loss and brain atrophy. In this condition, the measurement of ccf-mtDNA concentration configures as a potential biomarker for acute inflammatory stress. Whether this phenomenon is specific for MS or it rather reflects a generic neuro-inflammation still needs to be investigated. Since mitochondrial damage occurs in active MS lesions, mtDNA in the CSF could reflect its role as a DAMP. Considering mtDNA as a DAMP in MS, may explain the "inside-out theory" which suggests that inflammation is secondary to a primary intrinsic process within neurons or other cells such as oligodendrocytes. This neuro-immune concept consists in the formation of intracellular compounds, which trigger biochemical cascades leading to immunity activation (inflammasome) which once released from the cell recruit in turn a focal immune response. In this scenario, the "inside" mtDNA fragment would be the inflammatory stimulus, which clusters the intracellular cascade leading to a molecular complex, which triggers the immune response. Once such a complex is exposed "out" of the cell, immunity is strongly activated.

Thus, ccf-mtDNA may be a potential biomarker of cell death and non-specific tissue injury, and in the near future, it is supposed to become an innovative diagnostic tool in early stage screening and prognosis of several disorders.

ELIGIBILITY:
Inclusion Criteria:

• Clinical criteria for neurogenetic disease

Exclusion Criteria:

• absence of clinical condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: neurology analysis of patients by international trembling guidelines
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Neurology consulting | 1 week
  Radiological and neuro and physiological approces; different laboratory test (CSF analysis,ematological test);neurological impairment is assessed with Expanded Disability Status Scale and through radiological assessment, cognitive impairment.

SECONDARY OUTCOMES:
Molecular testing | 1 years
  Molecular analysis of ccf mtDNA
Cytokine measurements | 1 years
  The plasma levels of GM-CSF, IFN-γ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL- 8, IL-10, and TNF-α will be measured using the Human Cytokine Magnetic 10-Plex Panel (Thermo Fisher Scientific) according to the manufacturer's instructions. We will add the same plasma sample to each plate for cytokine multiplex assay and calculated inter assay CV (%). The quantization of plasma cytokines will be compared with the quantization of the ccf mtDNA and the clinical stage of the pathology
Statistical analyses. | 5 months
  Data will be presented as the mean ± standard deviation (SD). Categorical variables will compared using a chi-squared test. For a comparison of averages for the two groups, a Student's t-test will be used. When the data set will not normally distributed, a Mann-Whitney U-test will be used. Analysis of covariance (ANCOVA) controlling for age and sex will examined to evaluate the effects of age and sex on CFS, plasma or serum mtDNA copy number and cytokine levels. For a comparison of four groups, a one-way analysis of variance (ANOVA) followed by multiple comparisons with Tukey's method will used. Correlation coefficients between mtDNA copy number in plasma and cytokines will be calculated using Spearman's rank correlation coefficients. A P-value < 0.05 will considered as statistically significant and will corrected for multiple comparisons using Bonferroni's method.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Gambardella, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: Undecided